CLINICAL TRIAL: NCT03709550
Title: Phase Ib/II Study of Enzalutamide With Decitabine, a DNA Hypomethylating Agent, in Patients With Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Enzalutamide and Decitabine in Treating Patients With Metastatic Castration Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 51317; NCI-2018-01755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 51317 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Carcinoma Metastatic in the Bone; PSA Level Greater Than or Equal to Two; PSA Progression; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Decitabine; Injections; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (decitabine, enzalutamide) (Experimental): Participants receive decitabine IV over 1 hour on days 1-5 and enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Drug: Enzalutamide

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi

SUMMARY:
This phase I/II trial studies the side effects and best dose of decitabine and how well it works when given together with enzalutamide in treating patients with castration resistant prostate cancer that has spread to other places in the body. Androgen can cause the growth of prostate cancer cells. Drugs, such as enzalutamide, may lessen the amount of androgen made by the body. Decitabine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving decitabine and enzalutamide may work better in treating participants with castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of decitabine in combination with enzalutamide in patients with refractory metastatic castrate resistant prostate cancer (mCRPC). (Phase 1b) II. To determine the 12-month progression free survival rate of patients with enzalutamide-naive metastatic castrate resistant prostate cancer (mCRPC) treated with decitabine plus enzalutamide. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of decitabine in combination with enzalutamide in patients with refractory metastatic castrate resistant prostate cancer (mCRPC). (Phase 1b) II. To determine the overall response rate, overall survival and prostate specific antigen (PSA) changes in enzalutamide-naive mCRPC patients treated with decitabine plus enzalutamide. (Phase 2) III. To determine the safety and tolerability of decitabine in combination with enzalutamide in the study population. (Phase 2)

EXPLORATORY OBJECTIVES:

I. To determine the relationship between decitabine dose and plasma biomarkers (e.g., levels of HbF, LINE-1 methylation, number of circulating tumor cell's [CTC?s] and, NY-ESO expression in CTC?s). (Phase 1b) II. To explore plasma and tumor immune biomarkers associated with efficacy to the study combination. (Phase 2) III. To determine if treatment emergent neuroendocrine transformation is present as a result of the treatment combination of enzalutamide plus decitabine. (Phase 2) IV. Evaluate changes in stem cell reprogramming factors and deoxyribonucleic acid (DNA)/ribonucleic acid (RNA) markers resulting from the treatment combination. (Phase 2)

OUTLINE: This is a phase Ib, dose-escalation study of decitabine followed by a phase II study.

Participants receive decitabine intravenously (IV) over 1 hour on days 1-5 and enzalutamide orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of diagnosis of prostate cancer, all histological sub-types included.
* Documented progressive metastatic castrate resistant prostate cancer (mCRPC) based on at least one of the following criteria:

  * PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1week interval and a minimum PSA of 2 ng/mL
  * Soft-tissue progression defined as an increase >= 20% in the sum of the longest diameter (LD) of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions
  * Progression of bone disease (evaluable disease) or (new bone lesion[s]) by bone scan
  * If on an anti-androgen, must have documented progression 6 weeks after stopping anti-androgen therapy
* Willing to undergo a biopsy, if readily available biopsy site present, i.e., nodal or visceral metastasis (if adequate formalin-fixed, paraffin-embedded (FFPE) archival mCRPC samples are not available (or biopsy was taken longer than 6 months from start of study treatment), a fresh pre-treatment mCRPC biopsy needs to be obtained)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Have testosterone < 50 ng/dL. Note: Patients must continue primary androgen deprivation with an luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) if they have not undergone orchiectomy
* White blood cells >= 1.5 x 10^9/L (obtained within 14 days prior to treatment start)
* Platelets (UNVPLT) >= 100 x 10^9/L (obtained within 14 days prior to treatment start)
* Hemoglobin (HGB) >= 9 g/dL (obtained within 14 days prior to treatment start)
* Potassium (K), total calcium (CA) (corrected for serum albumin), magnesium, sodium (NA) and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication (obtained within 14 days prior to treatment start)
* International normalized ratio (INR) =< 1.5 (obtained within 14 days prior to treatment start)
* Serum creatinine (CREAT) =< 1.5 mg/dL or creatinine clearance > 50 mL/min (obtained within 14 days prior to treatment start)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN. If the patient has liver metastases, ALT and AST must still be =< 2.5 x ULN. Patients with liver metastases and AST/ALT above this limit will not be enrolled (obtained within 14 days prior to treatment start)
* Total serum bilirubin =< 1.5 x ULN; or total bilirubin (TBILI) =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert?s syndrome (obtained within 14 days prior to treatment start)
* Ability to swallow and retain oral medication (without crushing, dissolving or chewing tablets)
* Phase Ib only: Prior enzalutamide treatment and/or other approved treatments for CRPC are acceptable
* Phase II only: Participants MUST be treatment na?ve in the CRPC setting: i.e., no prior exposure to abiraterone acetate other specific CYP-17 inhibitors; no prior exposure to enzalutamide or investigational androgen receptor (AR) targeted agents; and no prior exposure to chemotherapy and or RAD-223
* Sexually active males must agree to use a condom during intercourse while taking the study drug and for at least 3 months after stopping study treatment. Sexually active males should not father a child during this period. A condom is required to be used by vasectomized men in order to prevent delivery of the drug via seminal fluid. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Phase II only: Prior exposure to abiraterone acetate
* Phase II only: Prior exposure to hypomethylating agents like azacytidine or decitabine
* Phase II only: Prior chemotherapy for castration resistant disease. Chemotherapy given in the castration-sensitive setting is permissible if stopped at least 4 weeks prior to treatment start
* Phase II only: Prior isotope therapy with strontium-89, samarium or radium-223 within 12 weeks of treatment start
* Participants with known symptomatic brain metastases
* Participant has a concurrent malignancy or malignancy within 3 years of treatment start, with the exception of adequately treated, basal or squamous cell carcinoma ornon-melanomatous skin cancer
* Participant has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory)
* Participant has clinically significant, uncontrolled heart disease and/or recent events including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to treatment start
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * On screening 12 lead electrocardiography (ECG), any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval > 109 msec or, Fridericia's correction formula (QTcF) > 450 msec. Congenital long QT syndrome or family history of long QT syndrome
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to treatment start:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids and pummelos, star-fruit and, Seville oranges
  * Medications that have a known risk to prolong the QT interval or induce Torsades de Pointes
  * Herbal preparations/medications, dietary supplements
* Patient who has received radiotherapy =< 4 weeks prior to start of treatment or limited field radiation for palliation =< 2 weeks prior to treatment start and, who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom >= 30% of the bone marrow was irradiated
* Patients with central nervous system (CNS) involvement
* Patients with seizure disorder
* Patient has not recovered from all toxicities related to prior anticancer therapies to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade < 1 (exception to this criterion: patients with any grade of alopecia are allowed to enter the study)
* Participant has any other concurrent severe and/or uncontrolled medical condition that would cause, in the investigator?s judgment, an unacceptable safety risk
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity determined by estimation of maximum tolerated dose assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Phase Ib) | Up to 28 days
  The dose level at which at least 2 out of 6 patients within the same cohort experience dose-limiting toxicity (DLT).
Incidence of adverse events assessed by NCI CTCAE version 4.03 (Phase Ib) | Up to 28 days after last dose
  Adverse event (AE) summaries will be organized by body system, frequency of occurrence, intensity (i.e., severity grade), and causality or attribution. Subjects who experience an AE more than once will be counted only once. The occurrence with the maximum severity will be used to calculate intensity. AEs deemed serious and those resulting in treatment withdrawal or death will be summarized separately.
Recommended phase II dose (Phase Ib) | Up to 28 days
Tumor response (Phase II) | Up to 24 months
  According to prostate specific antigen (PSA) response (longitudinally), Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, Prostate Cancer Working Group 3 (PCWG3) criteria and, a longitudinal mixed model for repeated measures of tumor burden: follow serial PSAs and follow target lesions on computed tomography scans and bone scans as per PCWG3 criteria.
Progression-free survival (PFS) (Phase II) | At 12 months
  The Kaplan-Meier product-limit estimator will be used to estimate PFS distributions.

OTHER OUTCOMES:
HbF measurements assessed by hemoglobin (Hgb) electrophoresis on peripheral blood (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Molecular pharmacodynamics assessed by flow cytometric assessment of DNMT1-protein in peripheral blood (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
LINE-1 methylation levels assessed in peripheral blood by pyrosequencing (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Number of circulating tumor cells (CTCs) and proportion of stem/progenitor cells in CTC population (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Presence or emergence of androgen receptor (AR) mutations, splice variants (ARv7), messenger ribonucleic acid (mRNA) levels in CTCs (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers. Correlation of gene expression levels will be measured using Pearson or Spearman correlation coefficients. Association of androgen profiles with clinical outcomes will use logistic regression or Cox proportional hazards regression, as appropriate.
Cancer-testis (CT) antigen, in particular NY-ESO-1 mRNA expression in CTCs (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers. Correlation of gene expression levels will be measured using Pearson or Spearman correlation coefficients.
Analyses of immune subsets (Phase II) | Up to 24 months
  Peripheral blood mononuclear cells (PBMC) will be assessed using multiparameter flow cytometry for immune subsets including but not necessarily limited to regulatory T cells (Tregs), myeloid-derived suppressor cell (MDSC), effector and exhausted CD4+ or CD8+ T-cells, and CD14+ monocytes. Assessment will include functional markers, i.e. PD-1, PD-L1, Tim-3, and CTLA-4. Will calculate the mean and standard deviation for these markers.
Evaluation of neuroendocrine lineage markers SYP, ASCL1, and CHGA (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Epigenetic reprogramming factors SOX2, EZH2, and DNMT1 assessed by biopsies (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Expression of luminal lineage markers like Androgen Receptor, KRT8 and KRT18 assessed in biopsies (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Decrease in DNMT1- protein level by > 50% (molecular pharmacodynamics) (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.
Analyses of immune signatures (Phase II) | Up to 24 months
  Will calculate the mean and standard deviation for these markers.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal Chatta, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States